CLINICAL TRIAL: NCT04254120
Title: Integrating Motivational Interviewing With Cognitive-behavioral Therapy for Anxiety Disorders, Depression, and Unhealthy Lifestyle Behaviors: a Feasibility Study
Brief Title: Integrating Motivational Interviewing With Cognitive-behavioral Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Benjamin Bohman, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KI-2013/1566-31/3
Record Dates: First submitted 2020-02-01; First posted 2020-02-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Anxiety Disorders and Symptoms; Depression; Life Style
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive-behavioral therapy (CBT) (Active Comparator)
  Interventions: Behavioral: Cognitive-behavioral therapy
- Integrated motivational interviewing and CBT (Experimental)
  Interventions: Behavioral: Integrated motivational interviewing and cognitive-behavioral therapy

INTERVENTIONS:
Behavioral: Cognitive-behavioral therapy — Psychological treatment focusing on changing cognitions and behaviors using information processing theory and learning theory approaches.
  Arms: Cognitive-behavioral therapy (CBT)
Behavioral: Integrated motivational interviewing and cognitive-behavioral therapy — Motivational interviewing is a psychological treatment approach focusing on increasing motivation by eliciting patient talk favoring behavior change and resolving patient ambivalence about change.
  Arms: Integrated motivational interviewing and CBT

SUMMARY:
Cognitive-behavioral therapy (CBT) is efficacious for anxiety disorders and depression, but not all patients achieve remission, and dropout is considerable. Motivational interviewing (MI) may strengthen motivation to change, and influence non-response and dropout. Research shows that MI as a pretreatment to CBT produces moderate effects compared to CBT alone. Studies integrating MI with CBT (MI-CBT) throughout treatment are scarce. The present study explored the feasibility of MI-CBT in routine psychiatric care, and compared CBT alone to MI-CBT for anxiety disorders, depression, and unhealthy lifestyle behaviors. The Anxiety, Depression, Diet, Alcohol, Physical activity, and Tobacco (ADDAPT) feasibility study had a randomized controlled design, and data were analyzed using hierarchical regression.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* A principal diagnosis according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) of panic disorder, social anxiety disorder, obsessive-compulsive disorder, generalized anxiety disorder, posttraumatic stress disorder, or major depressive disorder
* At least one of the following unhealthy lifestyle behaviors: unhealthy eating habits, hazardous use of alcohol, insufficient physical activity, or tobacco use, according to screening criteria suggested by the National Board of Health and Welfare

Exclusion Criteria:

* Psychotic symptoms
* DSM-IV-TR criteria for substance abuse other than alcohol
* DSM-IV-TR criteria for substance dependence including alcohol
* Moderate to severe suicide risk according to the Mini-International Neuropsychiatric Interview or a score of 2 or above on item 9 on the Patient Health Questionnaire 9
* Another simultaneous psychological treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2014-02-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
Index measure of aggregated psychiatric symptoms | 12 weeks
  Symptoms of principal anxiety disorder or principal depression, expressed as z scores; higher scores indicate more severe symptoms
Index measure of aggregated unhealthy lifestyle behaviors | 12 weeks
  Unhealthy lifestyle behaviors related to diet, physical activity, alcohol, or tobacco, expressed as z scores; higher scores indicate more problematic behaviors

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Bohman, Principal Investigator — Karolinska Institutet
Locations (1):
- WeMind Psykiatri AB, Stockholm, Sweden